CLINICAL TRIAL: NCT01783275
Title: The Effect of Exercise on Hepatic Glucose Metabolism in Type 2 Diabetes Mellitus
Brief Title: The Effect of Exercise on Hepatic Glucose Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Jason Winnick, Principal Investigator, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 121031; DK093799 (Other: NIDDK)
Record Dates: First submitted 2012-07-19; First posted 2013-02-04 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: Obesity; Type 2 diabetes; Liver
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise (Experimental): 12 weeks of aerobic exercise
  Interventions: Behavioral: Aerobic exercise
- Control (No Intervention): 12 weeks with no change in diet or exercise habits (weight maintenance).

INTERVENTIONS:
Behavioral: Aerobic exercise — 12 weeks of aerobic exercise with weight maintenance
  Arms: Aerobic Exercise

SUMMARY:
It is known that obesity and/or physical inactivity greatly increase a person's risk of developing heart disease and other serious health problems. This is partly because diabetes is associated with inflammation, oxidative stress, and insulin resistance. Diabetes is also associated with high levels of triglycerides in the blood and tissues such as the liver (known as fatty liver or steatosis). This elevation of fat in the liver is known to cause liver insulin resistance and impair the function of the liver and this impairment contributes to the development of diabetes.

Studies have shown that both aerobic exercise and weight loss have beneficial results on insulin resistance. However, the cause of this benefit remains unclear. We know that both aerobic exercise and/or weight loss can improve how muscle responds to insulin. However, it is also known that aerobic exercise and/or weight loss lowers liver fat content, thereby making it possible that the liver's response to insulin is also improved by weight loss and/or exercise training. An improved responsiveness of the liver to insulin could lower blood sugar levels after a meal and it could also lower morning blood sugar levels. However, very little is known about how exercise and/or weight loss improves liver function in people with type 2 diabetes.

Hypothesis 1: Improved hepatic insulin sensitivity, as a result of exercise training will increase the amount of glucose from an oral load that is taken up by the liver in subjects with DM.

Hypothesis 2: Increases in hepatic insulin sensitivity as a result of exercise will cause reductions in EGP during the fasted state, and will improve the suppression of EGP seen in response to hyperinsulinemia.

ELIGIBILITY:
Inclusion Criteria:

* 40-60 yrs of age
* sedentary lifestyle
* stable weight
* BMI 30 - 40kg/m2
* Hgb A1c <8.5
* Type 2 diabetes

Exclusion Criteria:

* Use of insulin
* Use of TZDs

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Splanchnic glucose uptake | 3 years
  Improved hepatic insulin sensitivity, as a result of lifestyle intervention, will increase the amount of glucose from an oral load that is taken up by the liver in subjects with DM.

SECONDARY OUTCOMES:
Endogenous glucose production | 3 years
  Increases in hepatic insulin sensitivity as a result of lifestyle intervention will cause reduced EGP during the fasted state, and in response to hyperinsulinemia.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Winnick, PhD, Principal Investigator — Vanderbilt University Medical Center; Naji Abumrad, MD, Study Chair — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No